CLINICAL TRIAL: NCT01233960
Title: A Multicenter, Open-label Study to Evaluate the Safety of PROCHYMAL® (Remestemcel-L) Intravenous Infusion in Subjects Who Have Received Previous Remestemcel-L Induction Treatment for Treatment-refractory Moderate-to-severe Crohn's Disease
Brief Title: Evaluation of PROCHYMAL® for Treatment-refractory Moderate-to-severe Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD 611
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2020-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Adult Stem Cell Therapy; inflammation of the gastrointestinal tract
MeSH Terms: conditions — Crohn Disease | interventions — remestemcel-l

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prochymal (Experimental): Infusions of Prochymal on days 42-45, 84-87, and 126-129 after first infusion in Protocol 603. Each infusion of PROCHYMAL (remestemcel-L) will contain 200 million cells.
  Interventions: Drug: adult human mesenchymal stem cells

INTERVENTIONS:
Drug: adult human mesenchymal stem cells — PROCHYMAL will be administered IV in a total volume of 300 ml (200 million cells) at a rate of 4-6 ml/minute. Treatments will be administered on Days 42-45, Days 84-87, and Days 126-129 following first infusion in Protocol 603.
  Other Names: Prochymal; remestemcel-L

SUMMARY:
To provide open-label re-treatment with PROCHYMAL to subjects enrolled in companion Protocol 603 to evaluate the safety in subjects with active Crohn's disease who are resistant to standard Crohn's disease therapies.

DETAILED DESCRIPTION:
Subjects will receive infusions of PROCHYMAL on Day 42, Day 84, and Day 126 after initial infusion of PROCHYMAL in Protocol 603. Each infusion will contain 200 million cells. As subjects will be required to be in Protocol 603 during the entire duration of their participation in Protocol 611, all concomitant medication and safety information will be monitored by Protocol 603 and the combination of data from the two protocols

ELIGIBILITY:
Inclusion Criteria:

* Subject must have qualified for, enrolled in, and provided written informed consent form (ICF) and authorization for use and disclosure of protected health information (PHI) for Protocol 603 after the August 3, 2010.
* Subject successfully completed all screening assessments in Protocol 603 as required by Protocol 603.
* Subject successfully completed the full course of each of the four infusions of investigational agent on Days 0, 3, 7, and 14 of Protocol 603 after August 3, 2010.
* Subject must enroll in Protocol 611 on or before the 45th day after first infusion in Protocol 603.
* Subject must provide written ICF and authorization for use and disclosure of PHI for Protocol 611.

Exclusion Criteria:

* Subject is unwilling or unable to adhere to requirements of Protocol 611.
* Subject had confirmed respiratory distress during a PROCHYMAL infusion in any prior PROCHYMAL study.
* Subject had a serious adverse event in any previous PROCHYMAL study that was deemed by the principal investigator of that study to be possibly or probably related to PROCHYMAL and also that was within 48 h after a PROCHYMAL infusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-11-29 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2014-09-15 (Actual)

PRIMARY OUTCOMES:
Disease remission | 180 Days after first infusion in Protocol 603
  Crohn's Disease Activity Index (CDAI) at or below 150 and increase in IBDQ

SECONDARY OUTCOMES:
Disease Improvement | 180 Days after first infusion in Protocol 603
  CDAI response to treatments is defined as a CDAI of 150 or below, or a reduction in CDAI of at least 100 points.
Improvement in Quality of Life (IBDQ) | 180 Days after first infusion in Protocol 603
  IBDQ response to treatment is defined as IBDQ of 170 or above, or an increase in IBDQ of at least 16 points.
Number of Adverse events as a measure of safety | 180 Days after first infusion in Protocol 603
Infusional toxicity as a measure of safety and tolerability | 180 Days after first infusion in Protocol 603
  Infusional toxicity will be evaluated by continuously monitoring the subject's vital signs and O2 saturation by pulse oximetry from the time of PROCHYMAL administration until two hours after infusion is complete.

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, Study Director — Mesoblast, Inc.
Locations (20):
- United States (16):
  - University of California, San Francisco, San Francisco, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - University of Chicago, Chicago, Illinois
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Saint Louis Center for Clinical Research, St Louis, Missouri
  - St. Louis Center for Clinical Studies, St Louis, Missouri
  - Dartmouth HItchcock Medical Center, Lebanon, New Hampshire
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Gastroenterology Center of the Midsouth, PC, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - McGuire Research Institute, Richmond, Virginia
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
- New Zealand (2):
  - University of Otago, Christchurch
  - Waikato Hospital, Hamilton